CLINICAL TRIAL: NCT01150708
Title: A Prospective Natural History Study of Patients With Syringomyelia
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100143; 10-N-0143
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-13

CONDITIONS: Syringomyelia; Arnold Chiari Deformity
Keywords: Syringomyelia; Magnetic Resonance Imaging; Natural History Study; Neurological Examination; Natural History
MeSH Terms: conditions — Syringomyelia; Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chiari 1 with syringomyelia: Chiari I malformation with syringomyelia.
- Chiari 1 without syringomyelia: A Chiari I Malformation without syringomyelia is defined as descent of the cerebellar tonsils > 5 mm below the foramen magnum 79 without associated syringomyelia.
- Syringomyelia without chiari: A syrinx or syringomyelia is defined as an intramedullary cyst that extends / length > 1spinal segment.

SUMMARY:
Background:

* Syringomyelia is a disorder in which a cyst (syrinx) forms within the spinal cord and causes spinal cord injury, with symptoms worsening over many years, including paralysis, loss of sensation, and chronic pain. Researchers are interested in obtaining more knowledge about how a syrinx forms in order to develop safer and more effective treatments for syringomyelia and related conditions.
* The goal of surgical treatment of syringomyelia is to eliminate the syrinx and prevent further spinal cord injury. In most patients, surgery results in the syrinx becoming smaller, but the effect of surgery on a patient s muscle strength, pain level, and overall function has not been studied over time. In addition, some individuals with syringomyelia or related conditions are not considered to be good candidates for surgery, and more information is needed about potential alternative treatments for these individuals.
* By recording more than 5 years of symptoms, muscle strength, general level of functioning, and magnetic resonance imaging (MRI) scan findings from individuals who receive standard treatment for syringomyelia, researchers can obtain more information about factors that influence its development, progression, and relief of symptoms.

Objectives:

- To conduct a 5-year natural history study of individuals with syringomyelia and related conditions.

Eligibility:

- Individuals at least 18 years of age who have syringomyelia or related conditions (including pre-syringomyelia or Chiari I malformation without syringomyelia).

Design:

* This study requires 7 outpatient visits to the National Institutes of Health Clinical Center: an initial visit; a visit 3 months later; and visits 1, 2, 3, 4, and 5 years after the initial visit. An additional 10 days of inpatient treatment and testing will be required if surgery is needed during the study.
* The following tests will be performed during this study:
* Medical history and physical examination, which may also determine eligibility for surgery
* Detailed neurological history and examination
* Blood and urine samples
* MRI scans: Participants will have 2 scans at the initial evaluation, 2 scans at the 3-month visit, and 1 scan every year for the following 5 years.
* Additional neurological and imaging tests if needed, including a lumbar puncture to collect spinal fluid, a myelogram (imaging study) of the spinal fluid, and a computed tomography scan of the skull and spine.
* Participants who are surgical candidates will have additional tests along with the surgery, including diagnostic studies (electrocardiogram and chest X-ray) before surgery and an MRI scan 1 week after surgery.

DETAILED DESCRIPTION:
OBJECTIVE

The natural history of patients who have syringomyelia has not been addressed in a prospective study. Present surgical treatment of patients with syringomyelia and neurologic deficit results in disease stabilization in many but not all patients, although objective improvement is less common. Delayed deterioration is not uncommon. The natural history of patients with syringomyelia and without a neurologic deficit or an associated lesion is also uncertain. By identifying factors that influence syringomyelia progression and that affect the response to surgical treatment, we can acquire knowledge that will enable us to provide more accurate recommendations to future patients with syringomyelia regarding optimal surgical or non-surgical treatment of their condition.

STUDY POPULATION

This study will enroll patients with syringomyelia and patients who are at risk of developing syringomyelia, including patients with Chiari I malformation and patients with presyringomyelia.

DESIGN

Prospective radiological and clinical data will be collected over a 5-year period from patients with syringomyelia and patients at risk of developing syringomyelia. Patients with syringomyelia and a neurological deficit will be considered to be surgical candidates. In this group, neurologic and radiographic outcomes in patients that undergo surgery will be compared to those in patients that refuse surgical treatment. Patients with syringomyelia but without neurological deficit will not be considered to be surgical candidates. In this group, initial neurologic and radiographic findings will be compared to those found one year after entrance into the study. Any patient with syringomyelia that develops progressive neurological deficit will be offered surgical treatment for his/her condition. In this study we will also prospectively collect information on processes that may influence the development and progression of syringomyelia, such as trauma and inflammatory diseases.

OUTCOME MEASURES

The primary outcome measure will be the change in motor strength, as measured by the American Spinal Injury (ASIA) Grading Scale, over 1 year. The secondary outcome measure will be the change in maximal syrinx diameter over 1 year in surgical candidates (surgically-treated vs. surgically untreated) and in non-surgical candidates.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this research study, the subject must:

1. Be 18 years of age or older.
2. Have syringomyelia, presyringomyelia, or Chiari I malformation without syringomyelia.
3. Be able to give informed consent.

ADDITIONAL CRITERIA FOR PATIENTS THAT MAY UNDERGO SURGERY (not required for study inclusion)

1. new or increased impairment in sensation, strength, or walking within the previous 2 years; and
2. an MRI-scan showing a syrinx or the presence of abnormal fluid and swelling in the spinal cord; the abnormality in the spinal cord must be located in a part of the spinal cord that could produce the patient s symptoms; and
3. evidence of abnormalities at the base of the skull or within the spine that are often associated with syringomyelia, or abnormalities in CSF circulation that increase the pressure of the cerebrospinal fluid; and
4. medical health that is sufficient to allow the subject to withstand a major surgical procedure and to remain active during the recovery period after surgery.

EXCLUSION CRITERIA:

The subject will not be eligible to participate in this research study if the subject:

1. Is pregnant (because multiple MRI scans might injure a fetus).
2. Cannot have an MRI scan as determined by the radiologist (see the risks below).
3. Has a problem with bleeding that cannot be corrected.

Note: Prior surgery for syringomyelia does not result in exclusion from the study if there is radiographic evidence of recurrent or persistent syringomyelia after surgery for this condition (failed previous surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is 180 patients with syringomyelia or with a condition that predisposes to the formation of syringomyelia such as presyringomyelia or Chiari I malformation without syringomyelia. A syrinx or syringomyelia is defined as an intramedullary cyst that extends / length > 1 spinal segment. Presyringomyelia will be defined as T2 hyperintensity > 4mm diameter extending over one spinal segment and associated with either Chiari I Malformation or a spinal lesion.A Chiari I Malformation without syringomyelia is defined as descent of the cerebellar tonsils > 5 mm below the foramen magnum without associated syringomyelia.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-08-03 (Actual)

PRIMARY OUTCOMES:
Change in ASIA Score | 1 year
  Patients with syringomyelia and a neurological deficit will be considered to be surgical candidates. In this group, neurologic and radiographic outcomes in patients that undergo surgery will be compared to neurologic and radiographic outcomes in patients that refuse surgical treatment. The primary outcome variable will be the change in motor strength in muscles of the upper and lower extremities as assessed by the American Spinal Injury (ASIA) Grading Scale. The change in ASIA score in patients between before surgery and one year after surgery will be compared to the one-year change in ASIA score in patients not receiving surgery (see Section 11, Statistical Analysis).

SECONDARY OUTCOMES:
Change in maximal Syrinx Anteroposterior Diameter | 1 year
  A secondary outcome measure will be the change in maximal syrinx anteroposterior diameter over 1 year in the surgical candidate group.Comparison will be made between groups that either undergo surgery or refuse surgical treatment. Another secondary outcome measure will be the change in maximal syrinx anteroposterior diameter over 1 year in the group of subjects that are not candidates for surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agarwalla PK, Dunn IF, Scott RM, Smith ER. Tethered cord syndrome. Neurosurg Clin N Am. 2007 Jul;18(3):531-47. doi: 10.1016/j.nec.2007.04.001. PMID 17678753
- [Background] Anderson NE, Willoughby EW, Wrightson P. The natural history of syringomyelia. Clin Exp Neurol. 1986;22:71-80. PMID 3581513
- [Background] Andrews BT, Weinstein PR, Rosenblum ML, Barbaro NM. Intradural arachnoid cysts of the spinal canal associated with intramedullary cysts. J Neurosurg. 1988 Apr;68(4):544-9. doi: 10.3171/jns.1988.68.4.0544. PMID 3280748
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-N-0143.html